CLINICAL TRIAL: NCT06754189
Title: Safety and Performance of UCon Patch Electrode for the Treatment of Overactive Bladder (OAB) and Bowel Dysfunction (BD) - A Pivotal Clinical Investigation
Brief Title: Safety and Performance of UCon Patch Electrode
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnoCon Medical (Industry)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK_PIVO_01
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Urge; Nocturia; Urinary Frequency More Than Once at Night; Urinary; Incontinence, Nighttime Urinary; Fecal Incontinence; Fecal Incontinence With Fecal Urgency
Keywords: Urinary Incontinence; Fecal Incontinence; Urge incontinence; Neurostimulation; Dorsal Genital Nerve
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Nocturia; Nocturnal Enuresis; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Participants are assigned to a treatment group and a sham group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Electrical stimulation (Time Limited stimulation) to the dorsal genital nerve.
  Interventions: Device: Time Limited stimulation
- Sham group (Sham Comparator): Sham stimulation to the dorsal genital nerve.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Time Limited stimulation — The participant self-administer 30 min. of electrical stimulation using Time Limited stimulation to the dorsal genital nerve (DGN) for 6 weeks using UCon with the UCon-Patch electrode.
  Other Names: UCon-Patch
  Arms: Treatment group
Device: Sham stimulation — The participant self-administer 30 min. of sham stimulation to the dorsal genital nerve (DGN) for 6 weeks using a sham device with the UCon-Patch electrode.
  Other Names: UCon-Sham
  Arms: Sham group

SUMMARY:
UCon is a medical device for treating the symptoms of overactive bladder (OAB) and bowel dysfunction (BD). It electrically stimulates the DGN through the skin to obtain modulated behavior of the bladder/bowel musculature e.g., suppressing undesired bladder/bowel activity to relieve the symptoms of the patient.

This pivotal clinical investigation is designed as a stratified-randomized, single-blinded, controlled, confirmatory, prospective, multicenter clinical investigation.

DETAILED DESCRIPTION:
The overall purpose of this pivotal clinical investigation is to evaluate the UCon device with a Patch Electrode with respect to clinical safety and device performance in a cohort of 180 patients with OAB/BD over a period of 12 weeks.

The participants participate in a 12-week intervention period. For weeks 1-6, participants will be randomized (2:1 randomization) to either a treatment group using UCon-Patch with Time Limited stimulation or a sham group using UCon-Sham with sham stimulation. Participants in the treatment group will receive the actual stimulation with the intent of improving their symptoms, whereas those in the sham group will receive sham stimulation for short periods of time believed not to be capable of improving their symptoms.

For weeks 7-12 of the intervention periods, the treatment group has the opportunity to add Urge stimulation to the Time Limited stimulation, while the sham group shifts to using UCon-Patch Time Limited stimulation.

To assess the safety and performance of the UCon device on equal terms with similar devices in the market, the full intervention period with UCon will be conducted over 12 weeks, evaluating safety aspects of UCon on longer terms and confirming continued effects after 6 weeks in the treatment group. Additional analyses on data related to primary and secondary endpoints with safety and performance data from the 12-week follow-up will also be performed, but the primary analysis will focus on baseline and 6-week follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 years of age.
* Participant is diagnosed with OAB or BD.
* Participant is able to consent, communicate, provide feedback, and understand and follow instructions in Danish during the course of the investigation, including operation of the device at home.

Exclusion Criteria:

* Participant has genital anatomy that does not allow for proper electrode placement or stimulation of the DGN.
* Participant has an active infection in the genital area, including skin infections.
* Participant has injured or irritated skin in the genital area, where the electrode is placed.
* Participant is medically unstable (acute illness or complication of a chronic condition, apart from the OAB or BD, that might affect the participant's participation in the investigation).
* Participant has an implanted pacemaker, implantable drug pump or other active medical devices (any medical device that uses electrical energy or other sources of power to make it function).
* Participant is pregnant, nursing, planning a pregnancy (to be confirmed with a negative pregnancy test) or has given birth within the previous 12 months. Women of childbearing potential must maintain effective contraception* during the clinical investigation.
* Participant is enrolled or planning to enroll in another conflicting clinical investigation or was enrolled in an investigational drug trial within the previous 12 weeks or medical device investigation within 12 weeks of enrolment.
* Participant has previously participated in a clinical investigation with UCon.
* Participant has failed (lack of effectiveness) other neuromodulation treatments, e.g. sacral neuromodulation (SNM) within the previous 2 years.
* Participant has a neurological disease, e.g., chronic inflammatory demyelinating polyneuropathy, multiple sclerosis, stroke, central nervous system (CNS) tumors, Parkinson´s, spinal cord injury, diabetic neuropathy, Guillain-Barré syndrome.
* Participant has a history of cancer in the pelvic region, is currently receiving cancer treatment, or has received radiation therapy in the pelvic region.
* Participant had surgery in the pelvic region within the previous 6 months. If it can be excluded that the participant's symptoms are related to the surgery, they can be included in the clinical investigation.
* Participant has addictive behavior defined as the abuse of alcohol, cannabis, opioids, or other intoxicating drugs.

  * The following contraception is considered effective: Intrauterine device, hormonal contraceptives such as birth control pills, implants, contraceptive patch, vaginal ring, and contraceptive injection.

Exclusion Criteria specific for OAB:

* Participant is planning or has a scheduled surgery/diagnostic procedure (within the duration of their participation) for any condition, that would require catheterization. Or have a prolonged hospitalization that would affect the ability to complete the stimulation.
* Participant (male) has symptoms of bladder outlet obstruction, e.g., caused by benign prostatic hyperplasia or prostate cancer.
* Participant has polyuria or symptoms of polyuria.
* Participant has a current or reoccurring urinary tract infection (≥3 or more within the previous 12 months or ≥2 within the previous 6 months).
* Participant has a primary diagnosis of stress urinary incontinence (SUI) or mixed incontinence with SUI likely to confound outcome measures.
* Participant has Bladder Pain Syndrome or interstitial cystitis.
* Participant has had botulinum toxin (BOTOX) treatment in the pelvic region within 9 months or has lasting benefit from BOTOX.
* Participant has failed (lack of effectiveness) BOTOX treatment within the previous 2 years.
* Participants who demonstrate detrusor overactivity on a urodynamic test can be included.
* Participant has used antimuscarinics or β3 agonists within 2 weeks.
* Participant has started oestrogen therapy within 3 months or are planning to stop therapy when enrolled in the clinical investigation.

Exclusion Criteria specific for BD:

* Participant is planning or has a scheduled surgery/diagnostic procedure (within the duration of their participation), for any condition, that would influence their bowel movements (e.g., injection of bulking agents, radiofrequency energy, or ligation of haemorrhoids). Or have a prolonged hospitalization that would affect the ability to complete the stimulation.
* Participant is currently being treated with antibiotics.
* Participant has a history of uncontrolled diarrhoea in the past 3 months (usual or most common stool type over the preceding 3 months of 7 on the Bristol Stool Form Scale).
* Participant has a history of severe constipation in the past 3 months (usual or most common stool type over the preceding 3 months of 1 on the Bristol Stool Form Scale).
* Participant has a history of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis). Participants with irritable bowel syndrome can be included in the clinical investigation.
* Participant has undergone major anorectal or bowel surgery or has ongoing anorectal or bowel conditions where primary surgery is considered the best, e.g., congenital anorectal malformation, bowel resection surgery, unrepaired rectovaginal fistula, chronic 4th degree anal sphincter laceration, full thickness rectal/anal prolapse. If it can be excluded that the participant's symptoms are related to any of the above surgeries/conditions, they can be included in the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse device effects (SADEs). | At 12 weeks.
  Number of SADEs.
Ratio of treatment change [performance] of OAB symptoms. | Change from baseline at 6 weeks.
  Percentage of participants using UCon-Patch, compared to participants using UCon-Sham, demonstrating at least a 50% reduction in Urinary Urgency (UU) voids (with or without Urgency Urinary Incontinence, UUI).
Ratio of treatment change [performance] of BD symptoms. | Change from baseline at 6 weeks.
  Percentage of participants using UCon-Patch, compared to participants using UCon-Sham, demonstrating at least a 50% reduction in Faecal Urgency (FU) episodes OR at least a 50% reduction in Faecal Incontinence (FI) episodes.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs). | At 12 weeks.
  Number of AEs.
Ratio of treatment change [performance] of Urgency Urinary Incontinence. | Change from baseline at 6 weeks.
  Percentage of participants using UCon-Patch, compared to participants using UCon-Sham, demonstrating at least a 50% reduction in Urgency Urinary Incontinence (UUI).
Self-reported quality of life measures as assessed by the International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life Module (ICIQ-OABqol) questionnaire. | Change from baseline at 6 weeks.
  The ICIQ-OABqol score of participants using UCon-Patch, compared to participants using UCon-Sham (scores can range from 0 to 100, with lower values indicating higher QoL).
Faecal Urgency (FU) episodes. | Change from baseline at 6 weeks.
  Mean reduction in number of Faecal Urgency (FU) episodes of participants using UCon-Patch, compared to participants using UCon-Sham.
Faecal Incontinence (FI) episodes. | Change from baseline at 6 weeks.
  Mean reduction in number of Faecal Incontinence (FI) episodes of participants using UCon-Patch, compared to participants using UCon-Sham.
Self-reported quality of life measures as assessed by the Rockwood Fecal Incontinence Quality of Life Scale (FIQL) questionnaire. | Change from baseline at 6 weeks.
  The FIQL score of participants using UCon-Patch, compared to participants using UCon-Sham (the scale consists of 4 scales, with each scale ranging from 1-5, with 1 indicating a lower functional QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christensen, MD, Principal Investigator — Palle Juul Jensens Boulevard 99 DK-8200 Aarhus N
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense